CLINICAL TRIAL: NCT02032576
Title: Predictors of the Response and Relapse/Recurrence After ECT for Depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Ching-Hua Lin, MD, PhD, Chief of Adult Psychiatry Department, Kaohsiung Kai-Suan Psychiatric Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSPH-2008-12
Record Dates: First submitted 2012-06-03; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Major Depressive Episode
Keywords: major depressive episode, electroconvulsive therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECT for depressed patients (Experimental): electroconvulsive therapy with a bipolar brief pulse square wave
  Interventions: Device: ECT for depressed patients

INTERVENTIONS:
Device: ECT for depressed patients — electroconvulsive therapy with a bipolar brief pulse square wave
  Other Names: bilateral ECT with a bipolar brief pulse square wave

SUMMARY:
Objective: Psychiatrists have long sought a quantifiable biomarker of electroconvulsive therapy (ECT) response. Although ECT is highly effective for treatment of patients with major depressive episode, a high rate of relapse/recurrence is a major problem after discontinuation of ECT. The purpose of this study is to examine the factors related to the response of ECT, to predict ECT response early, and to investigate the clinical predictors affecting the time to relapse/recurrence after ECT.

Methods: Patients with major depressive episode who require ECT treatment will be enrolled. ECT will be performed regularly. The 17-item Hamilton Rating Scale for Depression (HAMD-17) and other scales will be assessed before ECT, after every 10 days, till to an expected average of 50 days, and monthly during the 6-month follow-up period. Other measures also will be performed before the first ECT, at an expected average of 50 days, and at the end of follow-up period. Predictors of the response and relapse/recurrence after ECT and early prediction of ECT response will be obtained by statistic methods.

DETAILED DESCRIPTION:
Objective: Electroconvulsive therapy (ECT) is a safe and the most effective treatment for patients with major depressive episode, but the mechanism underlying the therapeutic action of this treatment is still unknown. Psychiatrists have long sought a quantifiable biomarker of ECT treatment response. Till now, no biomarker of ECT is used in clinical practice, but potential biomarkers that have been studied include brain-derived neurotrophic factor (BDNF), DNA polymorphism, RNA, electroencephalogram (EEG), auditory evoked potential (AEP), and cognitive function test. Although ECT is highly effective for treatment of major depressive episode, a high rate of relapse/recurrence is a major problem after discontinuation of ECT. The purpose of this study is to examine the factors related to the response of ECT for patients with major depressive episode, to predict the ECT response, and to investigate the clinical predictors affecting the time to relapse/recurrence after ECT.

Methods: Subjects with major depressive episode diagnosed according to DSM-IV criteria who require ECT treatment will be enrolled for study. ECT will be performed regularly using a brief-pulse, constant-current device. ECT will be given two or three times a week. The 17-item Hamilton Rating Scale for Depression (HAMD-17), Clinical Global Impression-severity (CGI-S), global assessment scale (GAF), UKU side effect rating scale and other scales will be assessed before ECT, after every 10 days, till to an expected average of 50 days, and monthly during the 6-month follow-up period. Response will be defined as a reduction of 60% or more of the HAMD-17 score after treatment. Other measures collected before ECT and at an expected average of 50 days include Zung's Depression Scale (SDS), Short-Form 36 (SF-36), Work and Social Adjustment Scale (WSAS), plasma BDNF level, auditory evoked potentials (AEP), electroencephalography (EEG), neuropsychological test, and RNA. After ECT, CGI-S, HAMD-17, GAF and WSAS are reexamined monthly for 6 months. The definition of relapse/recurrence will be readmission, a HAM-D-17 score at least 18, or a CGI-S score at least 4 during the follow-up period. A logistic regression model will be used to obtain the predictors for ECT response. To establish the early prediction of ECT response, receiver operating characteristic curve (ROC) will be used to determine the cutoff point. Possible predictors related to relapse/recurrence will be analyzed using the Cox proportional hazards regression model.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive disorder or bipolar depression
* Poor drug response
* Severity or urgency of illness

Exclusion Criteria:

* Subjects cannot write the imform consents
* Subjects with severe physical illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Predictors of ECT response | an expected average of 50 days after initiation of ECT
  Response will be defined as a reduction of 60% or more of the HAMD-17 score after treatment. Potential factors related to ECT response will be assayed. Early prediction model of response will be established.
Predictors of relapse/recurrence after ECT | After ECT, HAMD-17 will be assessed monthly until the relapse/recurrence of the major depressive episode during the 6-month follow-up period.
  The definition of relapse/recurrence of the major depressive episode will be readmission or a HAMD-17 score at least 18. Predictors (demographic and clinical variables) associated with time to relapse/recurrence during the 6-month follow-up period will be assayed using survival analysis.

SECONDARY OUTCOMES:
The changes of plasma brain-derived neurotrophic factor (BDNF) level after ECT | Prior to undergoing the first ECT and at an expected average of 50 days, plasma BDNF will be tested.
  The association between response and the change of BDNF will be examined.
The changes of cognitive functions after ECT | Neuropsychological test will be performed before the first ECT and at an expected average of 50 days.
  The impact of ECT on cognitive functions will be assayed.
Assessments of safety for general adverse events after ECT | UKU Side Effect Rating Scale will be assessed before ECT, after every 10 days, till to an expected average of 50 days.
  General adverse events were evaluated by a standardized the UKU Side Effect Rating Scale.
The changes of quality of life after ECT | Short-Form 36 (SF-36) will be examined before the first ECT and at an expected average of 50 days.
  The association between response and the change of SF-36 will be examined.
The changes of psychosocial functioning after ECT | Work and Social Adjustment Scale (WSAS) will be examined before the first ECT and at an expected average of 50 days.
  The association between response and the change of WSAS will be examined.
The changes of auditory evoked potentials (AEP) after ECT | Prior to undergoing the first ECT and at an expected average of 50 days, AEP will be tested.
  The association between response and the change of AEP will be examined.
The changes of electroencephalography (EEG) after ECT | Prior to undergoing the first ECT and at an expected average of 50 days, EEG will be tested.
  The impact of ECT on EEG will be assayed.
The changes of RNA after ECT | Prior to undergoing the first ECT and at an expected average of 50 days, RNA will be extracted from the blood.
  The association between response and the change of RNA will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hua Lin, M.D., Study Chair — Kai-Suan Psychiatric Hospital
Locations (1):
- Kai-Suan Psychiatric Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Result] Wahlund B, von Rosen D. ECT of major depressed patients in relation to biological and clinical variables: a brief overview. Neuropsychopharmacology. 2003 Jul;28 Suppl 1:S21-6. doi: 10.1038/sj.npp.1300135. PMID 12827140
- [Result] Bourgon LN, Kellner CH. Relapse of depression after ECT: a review. J ECT. 2000 Mar;16(1):19-31. doi: 10.1097/00124509-200003000-00003. PMID 10735328
- [Result] Marano CM, Phatak P, Vemulapalli UR, Sasan A, Nalbandyan MR, Ramanujam S, Soekadar S, Demosthenous M, Regenold WT. Increased plasma concentration of brain-derived neurotrophic factor with electroconvulsive therapy: a pilot study in patients with major depression. J Clin Psychiatry. 2007 Apr;68(4):512-7. doi: 10.4088/jcp.v68n0404. PMID 17474805